CLINICAL TRIAL: NCT03844802
Title: Effectiveness of Real or Placebo Dry Needling Combined With Therapeutic Exercise in Adults With Chronic Neck Pain
Brief Title: Effectiveness of Dry Needling in Chronic Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Junta de Andalucia (Other Government)
Responsible Party: Principal Investigator, Fernando Piña Pozo, Associate Professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dry Needling
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Neck Pain
Keywords: neck pain; randomized control trial; trigger points; dry needling; physical therapy; placebo; therapeutic exercise
MeSH Terms: conditions — Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The therapist in charge of the evaluation will remain unaware of participants' allocation group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Local dry needling and exercise (Experimental): The intervention protocol will combine a home-based neck and shoulder exercise program and the use of deep dry needling in the locus of active or latent myofascial trigger points of different neck-shoulder muscles. Patients will receive 1 dry needling session a week during 3 consecutive weeks (3 sessions in total). They will also undergo the neck exercise program at home during these three weeks, and for the next three months.
  Interventions: Other: Local Dry needling and exercise
- Distal dry needling and exercise (Active Comparator): The intervention protocol will combine a home-based neck and shoulder exercise program and the use of deep dry needling in distant area from the location of active or latent myofascial trigger points of different neck-shoulder muscles. Therefore, dry needling will be applied in the same muscle but at a remote site from the locus of the myofascial trigger point, and, therefore, without evoking local twitch responses. Patients will receive 1 dry needling session a week during 3 weeks (3 sessions in total). They will also undergo the neck exercise program at home during these three weeks, and for the next three months.
  Interventions: Other: Distal Dry needling and exercise
- Sham/placebo dry needling and exercise (Active Comparator): The intervention protocol will combine a home-based neck and shoulder exercise program and the use of deep dry needling in the locus of active or latent myofascial trigger points of different neck-shoulder muscles. Patients will receive 1 "placebo dry needling" session a week during 3 weeks (3 sessions in total). Therefore, participants in this group will receive simulated dry needling (with sham placebo needles, that will not actually penetrate the skin) in those neck muscles with active or latent myofascial trigger points. As formerly stated, the placebo needles evoke mechanical stimulation without piercing the skin; hence, patients experience a pressure sensation similar to that of a "real" needle.They will also undergo the neck exercise program at home during these three weeks, and for the next three months.
  Interventions: Other: Sham dry needling and exercise
- Neck Exercise (Active Comparator): The intervention protocol will consist only a home-based neck and shoulder exercise program. Participants in this group will be also assessed for the presence of active or latent myofascial trigger points in the neck-shoulder muscles. As in the other groups, they will be advised to carry out the exercise protocol for three weeks and the following three months.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Local Dry needling and exercise — Deep dry needling will be applied bilaterally in the locus of active or latent myofascial trigger points of several neck shoulder muscles (scalene muscles, levator scapulae, splenius cervicis, multifidus cervicis and upper trapezius). The presence of active or latent myofascial trigger points will be assessed according to the diagnostic procedures described by Travell and Simons. The dry needling intervention technique will be the fast in-fast out Hong technique, with a minimum of 3 to 6 local twitch responses to be elicited.
  Patients will perform a home based therapeutic neck exercises program.
  Arms: Local dry needling and exercise
Other: Distal Dry needling and exercise — Patients in this group will undergo deep dry needling at a remote spot from the locus of the myofascial trigger point. As a result no local twitch response should be elicited. As in the previous group, dry needling will be carried out in the same assessed muscles (scalene muscles, levator scapulae, splenius cervicis, multifidus cervicis and upper trapezius) with active or latent myofascial trigger points, according to the diagnostic procedures described by Travell and Simons. The intervention technique chosen for these participants will be to insert the needle in a location in the same muscle, but far away (at least 1 to 1.5 cm) from the location of the myofascial trigger point. Likewise, the needle will be inserted without the intention to evoke local twitch responses. Therefore, the entry and exit of the needle will be performed in a slower fashion.
  Patients will perform a home based therapeutic neck exercises program.
  Arms: Distal dry needling and exercise
Other: Sham dry needling and exercise — Patients in this group will undergo sham-placebo dry needling. For that purpose, placebo dry needling will be carried out in the same muscles previously described (scalene muscles, levator scapulae, splenius cervicis, multifidus cervicis and upper trapezius) with active or latent myofascial trigger points. The intervention technique will be carried out in the locus of the trigger point but using placebo needles. For this placebo group, a simulation needle procedure using a Dong Bang placebo needle, similar to the Streitberger needle, will be used. The placebo needles evoke mechanical stimulation without piercing the skin; hence, patients experience a pressure sensation similar to that of a "real" needle.
  Patients will perform a home based therapeutic neck exercises program.
  Arms: Sham/placebo dry needling and exercise
Other: Exercise — Patients will perform a home based therapeutic neck exercises program.
  Arms: Neck Exercise

SUMMARY:
Objectives: To investigate the effect of combining real or placebo dry needling with therapeutic exercise in self-reported pain, pressure pain sensitivity, neck disability, global rating of change (GROC) scale, muscle viscoelastic properties (muscle tone and stiffness) and left/right discrimination ability in adults with chronic non-specific neck pain.

Design: Quantitative, experimental, longitudinal, prospective, and single blinded study.

Subjects: Participants aged between 18 and 60 years, and with non specific neck pain of at least 3 months of evolution.

Methods: Participants will be randomly allocated in four groups: a) isolated use of a home based therapeutic exercise (TE) program (TE Group); b) combination of the exercise program and the use of deep dry needling (DN) in neck shoulder muscles with active or latent myofascial trigger points (MTrPs) in order to elicit local twitch responses (LTR) (TE + local DN Group); c) therapeutic exercise combined with DN applied distally from the muscle areas with MTrPs and, therefore, without, eliciting LTRs (TE + distal DN Group); and d) therapeutic exercise program combined with placebo DN (TE + placebo DN Group).

DETAILED DESCRIPTION:
All groups will be instructed by a physiotherapist in the performance of protocol of neck-shoulder exercises. This program will be carried out at home for at least three days a week during three months. The exercise protocol includes active mobilization, stretching and strengthening (concentric/eccentric, isotonic, and isometric) exercises. All participants will be given a booklet with a detailed description of every single exercise.

Those participants included in any of the DN groups will undergo 3 sessions of treatment (1 session per week during 3 consecutive weeks). In each session, the physiotherapist in charge of the intervention will assess the presence of active or latent MTrPs in severa neck shoulder muscles. The selected muscles have been previously described as having a higher prevalence of MTrPs in adults with chronic neck pain: a) scalene muscles; b) levator scapulae; c) splenius cervicis; d) cervical multifidus; and e) upper trapezius trapezius. The location of the trigger points will be carried out following the recommendations and guidelines described in the literature.

Those in the TE + local DN group will receive deep DN, using a fast-in fast-out technique, as described by Hong. The needle, once inserted in the muscle with a 10 to 20 mm depth, will be mobilized in a quick ascending and descending motion, in order to evoke the so-called LTRs. A minimum of 3 to 6 LTRs will be elicited in each muscle.

For patients in the TE + distal DN group, the deep DN intervention will be carried out in those muscles with MTrPs, but at a remote location from the MTrP area. The same evaluation and intervention protocol previously described for the TE + local DN group will be carried out. The main difference is that, in this group, DN will not elicit LTRs. Instead, DN will be applied at a minimum distance of 1-1.5 cm from the MTrP locus.

Finally, in the TE + placebo DN group, the therapeutic exercise program will be combined with DN using using a Dong Bang placebo needle, similar to the Streitberger placebo needle. These needles are designed with a retractable system. Therefore, these placebo needles evoke mechanical stimulation without piercing the skin; hence, patients experience a pressure sensation similar to that of a "real" needle.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-specific mechanical neck pain.
* Pain lasting for more than 3 months of duration.
* Self-reported pain higher than 3 in the Numeric Pain Rating Scale.
* Self-reported neck disability higher than 5 in the Neck Disability Index.

Exclusion Criteria:

* Absence of pain during passive neck rotation.
* Higher pain intensity in neutral position than during passive neck rotation.
* Absence of ipsilateral pain during passive neck rotation.
* Previous history of surgery of the cervical spine or upper extremity.
* Previous history of whiplash, diagnosis of fibromyalgia, or any neurological, inflammatory or rheumatological disease.
* Presence of two or more positive signs indicative of neural compression (sensitivity disorders, myotomic weakness in the upper extremities, or alteration in deep tendon reflexes).
* Radiological signs of root compression or spinal stenosis.
* Having received physical therapy treatment in the month prior to the start of the study.
* Analgesic and / or anti-inflammatory treatment in the last 72 h.
* Diagnosis of psychiatric disorders with ongoing medical treatment.
* Pregnancy or breastfeeding.
* Pending litigation in progress.
* Any contraindication to the use of dry needling.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Self-reported neck pain intensity in neutral head position at 6 months. | From Baseline to after treatment,with a 3-month and a 6- month follow up
  Current pain intensity in neutral head position, as assessed with a numeric pain rating scale (NPRS).The Numeric Pain Rating Scale is a 11-point rating scale that ranges from 0, which denotes no pain at all, to 10, which denotes the maximum bearable pain.
Change from baseline self-reported neck pain intensity associated to the most painful cervical rotation at 6 months | From Baseline to after treatment, with a 3-month and a 6- month follow up.
  Current pain intensity during the most painful passive cervical rotation, as assessed with a numeric pain rating scale (NPRS).The Numeric Pain Rating Scale is a 11-point rating scale that ranges from 0, which denotes no pain at all, to 10, which denotes the maximum bearable pain.
Change from baseline mean self-reported neck pain intensity during the last week at 6 months. | From Baseline to after treatment,with a 3-month and a 6- month follow up.
  The subject is asked about the mean pain intensity during the previous week, as assessed with a numeric pain rating scale (NPRS).The Numeric Pain Rating Scale is a 11-point rating scale that ranges from 0, which denotes no pain at all, to 10, which denotes the maximum bearable pain.
Change from baseline worst self-reported neck pain intensity in the last 24 hours at 6 months. | From Baseline to after treatment, with a 3-month and a 6- month follow up.
  The subject is asked about the highest neck pain intensity in the last 24 hours, as assessed with a numeric pain rating scale (NPRS).The subject is asked about theThe Numeric Pain Rating Scale is a 11-point rating scale that ranges from 0, which denotes no pain at all, to 10, which denotes the maximum bearable pain.

SECONDARY OUTCOMES:
Change from baseline self-reported neck related disability at 6 months. | From Baseline to after treatment, with a 3-month and a 6- month follow up.
  This will be assessed with the Neck disability index (NDI). The neck disability index is a condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. Each section is scored on a 0 to 5 rating scale, in which zero means no disability and 5 means the worst imaginable disability. The final score can range from 0 to 50 points (raw score) or from 0% to 100%, with 0 points or 0% denoting no activity limitations, and 50 points or 100% denoting complete activity limitation.
Change from baseline pressure pain sensitivity in neck shoulder muscles and brachial plexus nerve trunks at 6 months | From Baseline to after treatment, with a 3-month and a 6- month follow up.
  Pressure pain thresholds, defined as the minimum necessary pressure to evoke pain will be evaluated using a handheld electronic pressure algometer (model FPX 25, Wagner Instruments, Greenwich, CT, USA), with a 1-cm2 contact rubber probe. This outcome will be assessed over the upper trapezius, levator scapulae, anterior scalene and splenius cervicis muscles. The tibialis anterior muscle will be used as a remote location. Likewise, the pressure pain sensitivity will be evaluated over the median and cubital nerves.
Global Rating of Change. | After treatment, with a 3-month and a 6- month follow up.
  A 15-point numeral global rating of change scale will be used. This scale ranges from -7 (very much worse), through 0 (unchanged) to +7 (completely recovered). This is a patient self-reported scale that assesses whether the patient condition has gotten worse, better, or stayed the same. Participants are asked to quantify the magnitude of that change, whether positive or not.
Change from baseline muscle viscoelastic properties (muscle tone and stiffness) at 6 months | From Baseline to after treatment, with a 3-month and a 6- month follow up.
  The mechanical firmness of skeletal muscle in the absence of active contraction is related to the viscoelastic properties of the muscle tissue itself at rest, which can be quantified using myotonometry. The muscle tone and stiffness will be assessed over the upper trapezius, levator scapulae, anterior scalene, splenius cervicis and the tibialis anterior as a remote location. For this purpose, we will use a Myoton PRO (Myoton SA, Tallinn, Estonia) device. The MyotonPro is a low cost hand-held tool that uses multiple short impulses through a testing probe to measure several muscle properties, e.g., tone, stiffness, elasticity, and creep. The reliability and validity of the MyotonPro is well supported in healthy individuals, and in different musculoskeletal conditions.
Change from baseline left-Right discrimination ability at 6 months. | From Baseline to after treatment, with a 3-month and a 6- month follow up.
  The neck related left-right discrimination ability will be collected through the use of the Recognise app (2016 Noigroup, Adelaide, Australia, http://www.noigroup.com). We will use the app specific for the Neck version, using a Huawei P10 (5.15 "mobile phone, Huawei Technologies Co., Shenzhen, Guangdong.) Left / right discrimination can be defined as the process of identifying one side of the body as distinct from the other or identifying whether a part of the body is rotated to the left or right. We will assess both the accuracy and speed of discrimination.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto M Heredia-Rizo, PhD, Study Director — Physiotherapy Department, University of Sevilla, Spain; Fernando Piña-pozo, PT, Principal Investigator — Physiotherapy Department, University of Sevilla, Spain
Locations (1):
- University of Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: No